CLINICAL TRIAL: NCT01395836
Title: Management of New-Onset Postoperative Atrial Fibrillation Utilizing Insertable Cardiac Monitor Technology to Observe Recurrence of AF
Brief Title: Management of New-Onset Postoperative Atrial Fibrillation
Acronym: Monitor-AF
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Mikhael El Chami, Associate Professor, Emory University
Other Study IDs: IRB00047554a; EPEUHM (Other: Other)
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Atrial Fibrillation; Coronary Artery Disease; Post Operative Arrythmia
Keywords: Coronary Artery Bypass Grafting; Cardiology; Cardiac Electrophysiology; Cardiac Surgery
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Treatment: The "treatment" group will be medically managed based on data obtained from monthly transmissions of the implanted Cardiac Monitor.
- Control Group: The "control" group will be managed in the usual standard of care with physicians blinded to their ICM data.

SUMMARY:
One common occurrence following open heart surgery is an irregular rhythm from the top chambers of the heart known as atrial fibrillation (afib or AF). It is known that about 30% of patients who have had bypass surgery without having a heart valve replaced at the same time will develop AF. It is felt that this occurrence leads to factors that will affect a subjects health for the rest of their life. In studying this the investigators will see if post operative afib is an indicator of a person having afib and is not a condition that may only last during the post op recovery period as many physicians feel.The problem in question is, is post operative afib only transient or is it an indicator for more long term episodes of afib that may lead to other health concerns like stroke. Fifty subjects will be asked to participate. There will be to groups of 25 subjects. All subjects will have a device implanted under the skin that will be able to detect all types of heart rhythms. One group will get standard treatment and the physicians will be blinded to the recordings. The other group will be treated by the recording and the information about the amount of time in afib. The purpose of the study is to determine what the true occurrence of afib is for the first year after open heart surgery and to see if knowing this will alter the clinical management of this group of subjects.Currently most subjects are treated without knowing this information and based on that the arrhythmia will no longer happen after the heart is healed or recovered from the surgery. Most medications for controlling the heart rate and rhythm are stopped around 3 months. There is also a tendency to not to use blood thinning medications for the prevention of stroke after this time period. Stroke is one of the major complications from afib. Not all subjects are aware of the irregular heart beats so you can not depend on them to accurately know. They might feel episodes of very fast beating episodes or may become weak and fatigued. Weakness and fatigue are also normal during the first parts of recover from bypass surgery. By documenting the true episodes of afib the investigators can better understand if postoperative afib might need to be treated as a life long issue rather than a transient post operative issue. This treatment might change clinical management and decrease mortality.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able and willing to sign and date the Patient Consent Form.
* Subject is 18 years of age or older.
* Subject is expected to remain available for at least 12 months of follow- up visits.
* Subject is willing to comply with the protocol, including follow-up visits, medication compliance, carelink transmissions, and randomization assignment.
* Subject has a CHADS2 score of ≥ 1.
* Subject is hospitalized post isolated CABG or is within 72 hours post hospital discharge from a CABG procedure.
* Subject has no previous history of AF and has developed new-onset postoperative atrial fibrillation according to the established STS definition, which defines it as the occurrence of POAF or atrial flutter requiring treatment (i.e. beta-blockers, calcium-channel blockers, amiodarone, anticoagulation, or cardioversion).

Exclusion Criteria:

* Subject has a medically documented history of paroxysmal or persistent atrial fibrillation or atrial flutter.
* Subject is pregnant.
* Subject is enrolled or planning to participate in a concurrent drug and/or device study during the course of this study that would confound study results as determined by the study physician.
* Subject has previously or is scheduled to undergo valve repair or valve replacement during the course of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing isolated CABG at Emory University Hospital Midtown will be followed post-operatively and screened for inclusion to the trial.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2011-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The presence of AF at any post-operative points in time. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mikhael F El Chami, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital Midtown, Atlanta, Georgia, United States

REFERENCES:
- [Result] El-Chami MF, Merchant FM, Smith P, Levy M, Nelms AG, Merlino J, Puskas J, Leon AR. Management of New-Onset Postoperative Atrial Fibrillation Utilizing Insertable Cardiac Monitor Technology to Observe Recurrence of AF (MONITOR-AF). Pacing Clin Electrophysiol. 2016 Oct;39(10):1083-1089. doi: 10.1111/pace.12949. Epub 2016 Sep 22. PMID 27570120